CLINICAL TRIAL: NCT00385905
Title: Excel Drug-Eluting Stent Pilot Clinical Registry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Medical Systems Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2006-2
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

INTERVENTIONS:
Device: Excel Drug-eluting stent

SUMMARY:
The Trial aims to evaluate long-term efficiency of Excel stent in the inhibition of restenosis as well as the safety after the cessation of the 6-month anti-platelet drug treatment.

DETAILED DESCRIPTION:
30-day, 6-month, and 12-month clinical follow-up and 6 to 9-month IVUS or SCA follow-up to measure long-term efficiency of Excel stent in the inhibition of restenosis as well as the safety after the cessation of the 6-month anti-platelet drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who should fulfill with criteria of implanting Excel stents.
* Each patient enrolled is only allowed to implant Excel stents.
* Each patient are not allowed to be implanted more than 6 Excel stents.Also, 3 over-lapped stents are not allowed to be implanted in the same vessel(3-5mm overlapping needed; length of stents totally are not allowed to be over 80mm; fully post-dilated is essential for overlapping).
* Patients acknowlegement to the trial is essential.

Exclusion Criteria:

* AMI withine 1 week.
* Patients who do not suitable to Excel stenting.(For example, non-tolerant to anti-platelet drug or cardiac/non-cardiac surgery undergoing recently.)
* Patients who have multiple branch lesions can not apply single Excel stenting.
* Patients who refuse to sign the Trial Acknowledgement.
* Patients with intra-stent restenosis.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2006-02; Study Completion 2007-01

PRIMARY OUTCOMES:
12-month MACE

SECONDARY OUTCOMES:
30-day or 6-month MACE
6 to 9-month restenosis rate by SCA follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Ph.D., Study Chair — Shenyang Northern Hospital
Locations (1):
- Shenyang Nothern Hospital, Shenyang, Liaoning, China